CLINICAL TRIAL: NCT06837116
Title: Immunogenicity of an Intradermal Qdenga Vaccine Among Healthy Volunteers: A Pilot Study
Brief Title: Immunogenicity of an Intradermal Qdenga Vaccine Among Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sarunyou Chusri, Assoc. Prof. Sarunyou Chusri M.D. Ph.D., Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REC.67-475-14-1
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Dengue
Keywords: Safety; Immunogenicity; intradermal Qdenga
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SC ID (Active Comparator): subcutaneous Qdenga for 1st vaccination then intradermal Qdenga for 2nd vaccination
  Interventions: Biological: Vaccine
- SC SC (Active Comparator): subcutaneous Qdenga for 1st vaccination then subcutaneous Qdenga for 2nd vaccination
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Subcutaneous route vs Intradermal route

SUMMARY:
Official title: Immunogenicity of an intradermal Qdenga vaccine among healthy volunteers: A pilot study

DETAILED DESCRIPTION:
As in the setting of low- to middle-income countries, to demonstrating that lower doses of vaccine via intradermal route can still elicit robust immune responses, thereby lowering the overall cost of vaccination might be particularly meaningful ,with possible extra benefit of experiencing fewer side effects or risk of allergy. This study goal is to explores the potential of intradermal administration of Qdenga, hypothesizing that a lower dose via this route could achieve adequate immunogenicity compared to the standard subcutaneous administration, thus offering a cost-effective alternative particularly in low-resource settings where dengue is most prevalent.

ELIGIBILITY:
Inclusion Criteria:

* Thai adult aged 18-60 years, who not previously received dengue vaccine.
* The subjects are able to and willing to comply with the requirements of the clinical trial program and could complete the 3-month follow-up of the study.
* Individuals who are in good health condition at the time of entry into the trial as determined by medical history, physical examination and clinical judgment of the investigator and meet the requirements of immunization
* The subject can provide with informed consent and sign informed consent form

Exclusion Criteria:

* Have a medical history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* Be allergic to any component of the research vaccines or used to have a history of hypersensitivity or serious reactions to vaccination.
* Women with positive urine pregnancy test, pregnant or breast-feeding, or have a pregnancy plan within six months.
* Have acute infectious diseases, including dengue infection
* Have severe chronic diseases or condition in progress cannot be controlled. For example, poor controlled DM and uncontrolled HT.
* Have the history of urticaria 1 year before receiving the investigational vaccine.
* Have known underlying diseases of thrombocytopenia or other coagulation disorders (which may cause contraindications for intramuscular injection).
* Have needle sickness.
* Have the history of immunosuppressive therapy, cytotoxic therapy or systemic corticosteroids
* Have received blood products within 4 months before injection of investigational vaccines.
* Under anti-tuberculosis treatment.
* Not be able to follow the protocol, or not be able to understand the informed consent according to the researcher's judgment, due to various medical, psychological, social or other conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2025-04-19 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Prince of Songkla university, Hat Yai, Changwat Songkhla

IPD SHARING:
Plan to Share IPD: No
The data will be anonymized.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 adult volunteers were assessed for eligibility; 24 eligible participants were randomized into 2 groups (n = 12 per group).
Pre-assignment Details: 5 were excluded (4 have negative baseline dengue IgG, 1 withdraw from the study after randomization because of acute febrile illness prior to first dose vaccination).
Period: Overall Study
Arm/Group | SC ID | SC SC
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SC ID | SC SC | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 32.2 [23.9 to 40.5] | 39 [32 to 46] | 35.6 [27.3 to 43.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 2 | 1 | 3
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 21.18 [19.87 to 24.97] | 20.96 [20.34 to 23.34] | 21.05 [20.00 to 24.81]
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Dengue IgG Level
Description: To measure Antibody level for dengue by ELISA on day 0, day 30 and day 120 after 1st vaccination
Time Frame: Day 0 (Baseline), Day 30 (30 days post 1st vaccination) and Day 120 (30 days post 2nd vaccination)
Measure: Median (Inter-Quartile Range); unit: RU/ml
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
RU/ml
  Baseline | 108.9 [102.2 to 124.8] | 104.0 [104.0 to 113.0]
  Day 30 | 158.5 [151.1 to 164.5] | 143.2 [129.2 to 150.1]
  Day 120 | 148.6 [143.3 to 159.4] | 141.3 [127.1 to 152.8]
Statistical Analysis 1: Comparison: SC ID vs SC SC; Kruskal-Wallis test followed by Dunn's multiple comparisons test; Test type: Other; p < 0.01, Kruskal-Wallis; followed by Dunn's multiple comparisons test

2. Primary Outcome: CD4 T Cell Responses
Description: To measure T cell responses to dengue antigen by ELISpot on day 0, day 30 and day 120 after 1st vaccination.
Time Frame: Day 0 (Baseline), Day 30 (30 days post 1st vaccination) and Day 120 (30 days post 2nd vaccination)
Measure: Median (Inter-Quartile Range); unit: SFCs per 10^6 PBMCs
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
SFCs per 10^6 PBMCs
  Baseline | 22.0 [17.8 to 81.3] | 15.0 [5.0 to 38.0]
  Day 30 | 137.5 [60.8 to 178.3] | 103.0 [46.0 to 134.0]
  Day 120 | 98.5 [21.0 to 163.8] | 94.5 [67.3 to 127.0]

3. Primary Outcome: CD8 T Cell Response
Description: To measure T cell responses to dengue antigen by ELISpot on day 0, day 30 and day 120 after 1st vaccination.
Time Frame: Day 0 (Baseline), Day 30 (30 days post 1st vaccination) and Day 120 (30 days post 2nd vaccination)
Measure: Median (Inter-Quartile Range); unit: SFCs per 10^6 PBMCs
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
SFCs per 10^6 PBMCs
  Baseline | 5.0 [1.8 to 38.5] | 11.0 [1.0 to 47.0]
  Day 30 | 62.0 [24.5 to 105.5] | 11.0 [2.5 to 67.0]
  Day 120 | 6.0 [0.0 to 17.0] | 10.0 [2.5 to 49.5]

4. Secondary Outcome: All-Cause Mortality
Description: Death from any cause occurring from the first vaccination until the end of the 120-day follow-up period.
Time Frame: at day 7 and 30 post each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants
  All-Cause mortality | 0 | 0

5. Secondary Outcome: Serious Adverse Events
Description: Any untoward medical occurrence during the study period that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a congenital anomaly/birth defect, regardless of its relationship to the study vaccine.
Time Frame: at day 7 and 30 post each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

6. Secondary Outcome: Local Reactions
Description: - Include any reported pain, swelling, erythema or nodule at the vaccination site
Time Frame: at day 7 and 30 post each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 3 | 1

7. Secondary Outcome: Systemic Reactions
Description: fever, chill, fatique, headache, myalgia
Time Frame: at day 7 and 30 post each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 0 | 2

8. Secondary Outcome: Pain at Vaccination Site, 7 Day Post 1st Vaccination
Description: Injection-site pain reported during the 7-day period following the first vaccine dose.
Time Frame: 7 day post 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 2 | 1

9. Secondary Outcome: Erythema at Vaccination Site, 7 Day Post 1st Vaccination
Description: Erythema at vaccination site reported during the 7-day period following the first vaccine dose.
Time Frame: 7 day post 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 2 | 0

10. Secondary Outcome: Malaise, 7 Day Post 1st Vaccination
Description: Self-reported malaise during the 7-day period following the first vaccine dose.
Time Frame: 7 day post 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1

11. Secondary Outcome: Headache, 7 Day Post 1st Vaccination
Description: Self-reported headache during the 7-day period following the first vaccine dose.
Time Frame: 7 day post 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1

12. Secondary Outcome: Erythema at Vaccination Site, 7 Day Post 2nd Vaccination
Description: Erythema at vaccination site reported during the 7-day period following the second vaccine dose.
Time Frame: 7 day post 2nd vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | SC ID | SC SC
Number analyzed (Participants) | 12 | 12
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Day 37, 60 (7 and 30 days post 1st vaccination) and Day 97, 120 (7 and 30 days post 2nd vaccination)
Arm/Group | SC ID | SC SC
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SC ID (N=12) | SC SC (N=12)
Local reactions (Skin and subcutaneous tissue disorders) | 3 | 1 — pain, swelling, erythema or nodule
Systemic reactions (Immune system disorders) | 0 | 2 — Fever, chill, fatique, headache, myalgia
Pain at vaccination site, 7 day post 1st vaccination (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema at vaccination site, 7 day post 1st vaccination (Skin and subcutaneous tissue disorders) | 2 | 0
Malaise, 7 day post 1st vaccination (General disorders) | 0 | 1
Headache, 7 day post 1st vaccination (Nervous system disorders) | 0 | 1
Erythema at vaccination site, 7 day post 2nd vaccination (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This pilot study is limited by small sample size, short follow-up, and lack of neutralization assays and detailed T-cell phenotyping. These factors restrict interpretation of durability, serotype-specific responses, and immune correlates. Larger studies with extended immunologic assessments are planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT06837116/Prot_SAP_000.pdf